CLINICAL TRIAL: NCT02297230
Title: Locally Advanced Breast Cancer: Individualized Treatment Based On Tumor Molecular Characteristics
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI Left Institution prior to reaching accrual goal and analyzing data.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10289
Record Dates: First submitted 2014-10-27; First posted 2014-11-21 (Estimated); Results first posted 2018-01-18 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-09

CONDITIONS: Breast Cancer
Keywords: Locally Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy; Capecitabine; Trastuzumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1 Capecitabine and RT (Experimental): Her-2/neu negative patients will be given Capecitabine (xeloda, 750mg/m2 twice daily orally. Treatment should begin on day 1 of radiation therapy. The two doses should be taken about 30 minutes after eating (eg. after breakfast and after dinner). Treatment will be given for 10 weeks (for 6 weeks during radiation and for 4 weeks after radiation).
  Interventions: Radiation: Radiation Therapy (RT); Drug: Capecitabine
- Arm 2 Paclitaxel/Trastuzumab and RT (Experimental): Trastuzumab (Herceptin®) will begin on day 1 of radiation therapy and be administered weekly to Her-2/neu Positive patients. The first dose will be 4mg/kg given IV over 90 minutes. Weekly doses will be 2 mg/kg/week IV over 30 minutes.Paclitaxel 30 mg/m2 twice per week given IV over 1 hour.
  Interventions: Radiation: Radiation Therapy (RT); Drug: Trastuzumab; Drug: Paclitaxel
- Arm 3: Paclitaxel and RT (Experimental): Paclitaxel 30 mg/m2 twice per week given IV over 1 hour to Her-2/neu negative patients. Treatment will be initiated during the first week of radiation therapy and should be administered on a Monday/Thursday or Tuesday/Friday schedule.
  Interventions: Radiation: Radiation Therapy (RT); Drug: Paclitaxel
- Arm 4: Paclitaxel/Trastuzumab and RT (Experimental): Trastuzumab (Herceptin®) tx will be administered weekly, together with one of the 2 weekly doses of Paclitaxel to Her-2/neu Positive patients. The 1st dose will be 4mg/kg given IV over 90 minutes. Weekly doses will b given at a dose of 2 17mg/kg/week IV over 30 minutes. The Tx with Trastuzumab will continue weekly after the completion of the radiation tx until surgery & thereafter as per std of care up to 1 yr post surgery.Paclitaxel 30 mg/m2 twice per week given IV over 1 hour. Tx will be administered on a Monday/Thursday or Tuesday/Friday schedule.The radiation treatment will start within 1 week from the first dose of paclitaxel and trastuzumab.
  Interventions: Radiation: Radiation Therapy (RT); Drug: Trastuzumab; Drug: Paclitaxel

INTERVENTIONS:
Radiation: Radiation Therapy (RT) — Concurrent RT (to start within one week from first dose of Paclitaxel/Trastuzumab) to breast, supraclavicular, axillary fields, 45 Gy @ 1.8 Gy/fraction, + 14 Gy @ 2 Gy/fraction to the primary tumor. At the end of chemo-radiation, Trastuzumab will be continued weekly until surgery and as per standard of care after surgery for up to 1 year total.
Drug: Capecitabine — Capecitabine (Xeloda®) 750 mg/m2 twice/daily given orally. Treatment should begin on day 1 of radiation therapy. The two doses should be taken about 30 minutes after eating (eg. after breakfast and after dinner). Treatment will be given for 10 weeks (for 6 weeks during radiation and for 4 weeks after radiation).
  Other Names: Xeloda
  Arms: Arm 1 Capecitabine and RT
Drug: Trastuzumab — Trastuzumab (Herceptin®) treatment will be administered weekly, together with one of the two weekly doses of Paclitaxel. The first dose will be 4mg/kg given IV over 90 minutes. Subsequent weekly doses will be given at a dose of 2 mg/kg/week IV over 30 minutes. The treatment with Trastuzumab will continue weekly after the completion of the radiation treatment until surgery and thereafter as per standard of care up to 1 year post surgery.
  Other Names: Herceptin
  Arms: Arm 2 Paclitaxel/Trastuzumab and RT; Arm 4: Paclitaxel/Trastuzumab and RT
Drug: Paclitaxel — Paclitaxel 30 mg/m2 twice per week given IV over 1 hour. Treatment will be administered on a Monday/Thursday or Tuesday/Friday schedule.The radiation treatment will start within 1 week from the first dose of paclitaxel and trastuzumab. Pre-meds for paclitaxel should be based on the institutional standards; it is suggested that dexamethasone (Decadron®), 20 mg IV, be given with the first paclitaxel dose. If the patient tolerates the treatment, the dexamethasone may be tapered and/or discontinued for subsequent doses. Treatment will be given for 10 weeks (for 6 weeks during radiation and for 4 weeks following radiation).
  Other Names: Taxol
  Arms: Arm 2 Paclitaxel/Trastuzumab and RT; Arm 3: Paclitaxel and RT; Arm 4: Paclitaxel/Trastuzumab and RT

SUMMARY:
Paclitaxel 30 mg/m2 twice/week Trastuzumab 4mg/kg, loading dose, then 2 mg/kg weekly and Concurrent RT (to start within one week from first dose of Paclitaxel/Trastuzumab) to breast, supraclavicular, axillary fields, 45 Gy @ 1.8 Gy/fraction, + 14 Gy @ 2 Gy/fraction to the primary tumor. At the end of chemo-radiation, Trastuzumab will be continued weekly until surgery and as per standard of care after surgery for up to 1 year total.

**Surgery: Patients will undergo lumpectomy and axillary node dissection or modified radical mastectomy within two months following discontinuation of pre-operative systemic therapy, contingent upon recovery of skin toxicity. Pathologic response will be evaluated at the time of surgery. Additional tissue samples will be collected from the surgical specimen for assessment of tumor molecular characteristics.

***All patients may undergo four cycles of post-operative Standard AC (doxorubicin 60 mg/m2, cyclophosphamide 600 mg/m2) or four cycles of post-operative epirubicin and Cyclophosphamide (epirubicin 100 mg/m2, cyclophosphamide 600 mg/m2) if doxorubicin is not available Tamoxifen as well or any alternative antihormonal therapy may be prescribed for five years for patients with hormone receptor positive tumors. Herceptin (Trastuzumab) will be prescribed for a total of 1 year since first dose as per standard of care.

DETAILED DESCRIPTION:
Locally Advanced Breast Cancer: T greater than 3.0 cm. HER-2/neu positive. Patients with ipsilateral supraclavicular nodes are eligible. Patients with inflammatory breast cancer or distant metastases are excluded. Patients with prior treatment for their breast cancer are excluded. Patients must have adequate laboratory parameters and normal cardiac function. Patients receive Concurrent Radiation therapy with either Capecitabine, Paclitaxel and Herceptin. Capecitabine (Xeloda®) 750 mg/m2 twice/daily given orally. Treatment should begin on day 1 of radiation therapy. The two doses should be taken about 30 minutes after eating (eg. after breakfast and after dinner). Treatment will be given for 10 weeks (for 6 weeks during radiation and for 4 weeks after radiation).Trastuzumab (Herceptin®) will begin on day 1 of radiation therapy and be administered weekly. The first dose will be 4mg/kg given IV over 90 minutes. Subsequent weekly doses will be 2 mg/kg/week IV over 30 minutes. Paclitaxel 30 mg/m2 twice per week given IV over 1 hour. Treatment will be initiated during the first week of radiation therapy and should be administered on a Monday/Thursday or Tuesday/Friday schedule.Paclitaxel 30 mg/m2 twice per week given IV over 1 hour. Treatment will be initiated during the first week of radiation therapy and should be administered on a Monday/Thursday or Tuesday/Friday schedule.Trastuzumab (Herceptin®) treatment will be administered weekly, together with one of the two weekly doses of Paclitaxel. The first dose will be 4mg/kg given IV over 90 minutes. Subsequent weekly doses will be given at a dose of 2 mg/kg/week IV over 30 minutes. The treatment with Trastuzumab will continue weekly after the completion of the radiation treatment until surgery and thereafter as per standard of care up to 1 year post surgery.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven locally advanced breast cancer: STAGE IIB (T must be > 3.0 cm, N0), IIIA (T0N2, T1N2, T2N2, T3N1), IIIB (T4N0-2).
* HER-2/neu positive ( DAKO 3+ by Immunohistochemistry or FISH positive if Dako 2+)
* Metastatic breast cancer: limited to the subset of patients with intact breast, locally advanced tumor and involved ipsilateral supraclavicular nodes.
* Measurable disease required according to the RECIST criteria (Response Evaluation Criteria in Solid Tumors)
* Adequate laboratory values:
* Hgb > 10
* ANC(Absolute Neutrophil Count) > 1500
* Platelets > 150,000
* Cr < 1.5
* Liver function < 3 X normal.
* Patient > 18 years of age.
* Medically and psychologically able to comply with all study requirements.
* ECOG (Eastern cooperative Oncology group) performance score 0-1.
* Signed informed consent.

Exclusion Criteria:

* Stage 0, Stage I, Stage IIA.
* Previous XRT(Radiation therapy) or chemotherapy.
* Presence of distant metastases documented clinically or radiographically with the exception of ipsilateral supraclavicular nodes.
* Inflammatory breast cancer.
* Prior unanticipated severe reaction to fluoropyrimidine therapy or known hypersensitivity to 5-fluorouracil.
* Exclude pregnant or lactating woman.
* Woman of childbearing potential with either a positive or no pregnancy test at baseline.
* Woman of childbearing potential not using a reliable and appropriate contraceptive method.
* (Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential).
* Patient will agree to continue contraception for 30 days from the date of the last study drug administration.
* Serious concurrent infections.
* Clinically significant cardiac disease not well controlled with medication (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias ) or myocardial infarction within the last 12 months.
* Patients who have had an organ allograft.
* Patients with severe renal impairment (creatinine clearance below 30 mL/min [Cockcroft and Gault43]). In patients with moderate renal impairment (creatinine clearance 30-50 mL/min [Cockcroft and Gault43]) at baseline, a dose reduction to 75% of the XELODA starting dose is recommended. In patients with mild renal impairment (creatinine clearance 51-80 mL/min) no adjustment in starting dose is recommended.
* In phase I studies, those with any abnormal renal function, since toxicity will likely be affected by the presence of any significant renal dysfunction.
* Cockcroft and Gault Equation:
* (140 - age [yrs]) (body wt [kg])
* Creatinine clearance for males = --------------
* (72) (serum creatinine [mg/dL])
* Creatinine clearance for females = 0.85 x male value

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2002-06; Primary Completion 2014-12-02 (Actual); Study Completion 2014-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia C Formenti, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 Capecitabine and RT: Her-2/neu negative patients will be given Capecitabine (xeloda, 750mg/m2 twice daily orally. Treatment should begin on day 1 of radiation therapy. The two doses should be taken about 30 minutes after eating (eg. after breakfast and after dinner). Treatment will be given for 10 weeks (for 6 weeks during radiation and for 4 weeks after radiation).
  radiation therapy: Concurrent RT (to start within one week from first dose of Paclitaxel/Trastuzumab) to breast, supraclavicular, axillary fields, 45 Gy @ 1.8 Gy/fraction, + 14 Gy @ 2 Gy/fraction to the primary tumor. At the end of chemo-radiation, Trastuzumab will be continued weekly until surgery and as per standard of care after surgery for up to 1 year total.
  Capecitabine: Capecitabine (Xeloda®) 750 mg/m2 twice/daily given orally. Treatment should begin on day 1 of radiation therapy. The two doses should be taken about 30 minutes after eating (eg. after breakfast and after dinner). Treatment will be given for 10 weeks (for 6 weeks
- Arm 2 Paclitaxel/Trastuzumab and RT: Trastuzumab (Herceptin®) will begin on day 1 of radiation therapy and be administered weekly to Her-2/neu Positive patients. The first dose will be 4mg/kg given IV over 90 minutes. Weekly doses will be 2 mg/kg/week IV over 30 minutes.Paclitaxel 30 mg/m2 twice per week given IV over 1 hour.
  radiation therapy: Concurrent RT (to start within one week from first dose of Paclitaxel/Trastuzumab) to breast, supraclavicular, axillary fields, 45 Gy @ 1.8 Gy/fraction, + 14 Gy @ 2 Gy/fraction to the primary tumor. At the end of chemo-radiation, Trastuzumab will be continued weekly until surgery and as per standard of care after surgery for up to 1 year total.
  Trastuzumab: Trastuzumab (Herceptin®) treatment will be administered weekly, together with one of the two weekly doses of Paclitaxel. The first dose will be 4mg/kg given IV over 90 minutes. Subsequent weekly doses will be given at a dose of 2 mg/kg/week IV over 30 minutes. The treatment with Trastuzumab will continue weekly after the
- Arm 3: Paclitaxel and RT: Paclitaxel: Paclitaxel 30 mg/m2 twice per week given IV over 1 hour. Treatment will be administered on a Monday/Thursday or Tuesday/Friday schedule.The radiation treatment will start within 1 week from the first dose of paclitaxel and trastuzumab. Pre-meds for paclitaxel should be based on the institutional standards; it is suggested that dexamethasone (Decadron®), 20 mg IV, be given with
Period: Overall Study
Arm/Group | Arm 1 Capecitabine and RT | Arm 2 Paclitaxel/Trastuzumab and RT | Arm 3: Paclitaxel and RT | Arm 4: Paclitaxel/Trastuzumab and RT
Started | 11 | 11 | 11 | 11
Completed | 11 | 11 | 11 | 11
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm 2 Paclitaxel/Trastuzumab and RT: Trastuzumab (Herceptin®) will begin on day 1 of radiation therapy and be administered weekly to Her-2/neu Positive patients. The first dose will be 4mg/kg given IV over 90 minutes. Weekly doses will be 2 mg/kg/week IV over 30 minutes.Paclitaxel 30 mg/m2 twice per week given IV over 1 hour.
  r
- Total: Total of all reporting groups
Arm/Group | Arm 1 Capecitabine and RT | Arm 2 Paclitaxel/Trastuzumab and RT | Arm 3: Paclitaxel and RT | Arm 4: Paclitaxel/Trastuzumab and RT | Total
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 40
  >=65 years | 1 | 1 | 1 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 11 | 11 | 44
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 11 | 11 | 11 | 44

OUTCOME MEASURES:

1. Primary Outcome: Feasibility & Efficacy of Chemo-radiation While Targeting Treatment, Based on: Original Tumor Characteristics; to be Followed by [Need for] Conventional Post-operative Chemotherapy
Time Frame: 12/2014 (up to 12 years)
Population: Data were not collected as PI left institution prior to enrollment completion. PI terminated protocol.
Arm/Group | Arm 1 Capecitabine and RT | Arm 2 Paclitaxel/Trastuzumab and RT | Arm 3: Paclitaxel and RT | Arm 4: Paclitaxel/Trastuzumab and RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: To Assess the Pathological Response Rate and Compare it to That Achieved in Our Previous Phase I-II Trials of Concurrent Chemo-radiation.
Description: No data displayed because Outcome Measure has zero total participants analyzed.
Time Frame: 12/2014 (up to 12 years)
Population: Planned Statistical analysis was not performed for this secondary outcome measure. Study Terminated prematurely; PI left institution;
Groups:
- Arm 3: Paclitaxel and RT: Paclitaxel 30 mg/m2 twice per week given IV over 1 hour to Her-2/neu negative patients. Treatment will be initiated during the first week of radiation therapy and should be administered on a Monday/Thursday or Tuesday/Friday schedule.
  Concurrent RT (to start within one week from first dose of Paclitaxel/Trastuzumab) to breast, supraclavicular, axillary fields, 45 Gy @ 1.8 Gy/fraction, + 14 Gy @ 2 Gy/fraction to the primary tumor. At the end of chemo-radiation, Trastuzumab will be continued weekly until surgery and as per standard of care after surgery for up to 1 year total.
- Arm 4: Paclitaxel/Trastuzumab and RT: Trastuzumab (Herceptin®) tx will be administered weekly, together with one of the 2 weekly doses of Paclitaxel to Her-2/neu Positive patients.
  Concurrent RT (to start within one week from first dose of Paclitaxel/Trastuzumab) to breast, supraclavicular, axillary fields, 45 Gy @ 1.8 Gy/fraction, + 14 Gy @ 2 Gy/fraction to the primary tumor. At the end of chemo-radiation, Trastuzumab will be continued weekly until surgery and as per standard of care after surger
Arm/Group | Arm 1 Capecitabine and RT | Arm 2 Paclitaxel/Trastuzumab and RT | Arm 3: Paclitaxel and RT | Arm 4: Paclitaxel/Trastuzumab and RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: To Store Core Biopsies of the Original Tumor Before and After Treatment (From the Surgical Specimen) for Future Molecular Biology Studies in LABC.
Description: No data displayed because Outcome Measure has zero total participants analyzed.
Time Frame: 12/2014 (up to 12 years)
Population: Data were not collected as PI left institution prior to enrollment completion. PI terminated protocol.
Groups:
- Arm 1 Capecitabine and RT: radiation therapy: Concurrent RT (to start within one week from first dose of Paclitaxel/Trastuzumab) to breast, supraclavicular, axillary fields, 45 Gy @ 1.8 Gy/fraction, + 14 Gy @ 2 Gy/fraction to the primary tumor. At the end of chemo-radiation, Trastuzumab will be continued weekly until surgery and as per standard of care after surgery for up to 1 year total.
  Capecitabine: Capecitabine (Xeloda®) 750 mg/m2 twice/daily given orally. Treatment should begin on day 1 of radiation therapy. The two doses should be taken about 30 minutes after eating (eg. after breakfast and after dinner). Treatment will be given for 10 weeks (for 6 weeks during radiation and for 4 weeks after radiation).
- Arm 2 Paclitaxel/Trastuzumab and RT: Trastuzumab (Herceptin®) will begin on day 1 of radiation therapy and be administered weekly to Her-2/neu Positive patients. The first dose will be 4mg/kg given IV over 90 minutes. Weekly doses will be 2 mg/kg/week IV over 30 minutes.Paclitaxel 30 mg/m2 twice per week given IV over 1 hour.
  radiation therapy: Concurrent RT (to start within one week from first dose of Paclitaxel/Trastuzumab) to breast, supraclavicular, axillary fields, 45 Gy @ 1.8 Gy/fraction, + 14 Gy @ 2 Gy/fraction to the primary tumor
  Trastuzumab: Trastuzumab (Herceptin®) treatment will be administered weekly, together with one of the two weekly doses of Paclitaxel.
  Paclitaxel: Paclitaxel 30 mg/m2 twice per week given IV over 1 hour.
- Arm 3: Paclitaxel and RT: Paclitaxel 30 mg/m2 twice per week given IV over 1 hour to Her-2/neu negative patients. -
  radiation therapy: Concurrent RT (to start within one week from first dose of Paclitaxel/Trastuzumab) to breast, supraclavicular, axillary fields, 45 Gy @ 1.8 Gy/fraction, + 14 Gy @ 2 Gy/fraction to the primary tumor. At the end of chemo-radiation, Trastuzumab will be continued weekly until surgery and as per standard of care after surgery for up to 1 year total.
  Paclitaxel: Paclitaxel 30 mg/m2 twice per week given IV over 1 hour. Treatment will be administered on a Monday/Thursday or Tuesday/Friday schedule.The radiation treatment will start within 1 week from the first dose of paclitaxel and trastuzumab. Pre-meds for paclitaxel should be based on the institutional standards; it is suggested that dexamethasone (Decadron®), 20 mg IV, be given with
- Arm 4: Paclitaxel/Trastuzumab and RT: Trastuzumab (Herceptin®) tx will be administered weekly, together with one of the 2 weekly doses of Paclitaxel to Her-2/neu Positive patients. The 1st dose will be 4mg/kg given IV over 90 minutes. Weekly doses will b given at a dose of 2 17mg/kg/week IV over 30 minutes. The Tx with Trastuzumab will continue weekly after the completion of the radiation tx until surgery & thereafter as per std of care up to 1 yr post surgery.Paclitaxel 30 mg/m2 twice per week given IV over 1 hour. Tx will be administered on a Monday/Thursday or Tuesday/Friday schedule.The radiation treatment will start within 1 week from the first dose of paclitaxel and trastuzumab.
  radiation therapy: Concurrent RT (to start within one week from first dose of Paclitaxel/Trastuzumab) to breast, supraclavicular, axillary fields, 45 Gy @ 1.8 Gy/fraction, + 14 Gy @ 2 Gy/fraction to the primary tumor.
Arm/Group | Arm 1 Capecitabine and RT | Arm 2 Paclitaxel/Trastuzumab and RT | Arm 3: Paclitaxel and RT | Arm 4: Paclitaxel/Trastuzumab and RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: To Acquire Descriptive Information on Patient Adherence to Therapy and on Quality of Life During Treatment.
Description: Data were not collected as PI left institution prior to enrollment completion. Planned Statistical analysis was not performed for this secondary outcome measure.
Time Frame: 12/2014 (up to 12 years)
Population: No data displayed because Outcome Measure has zero total participants analyzed.
Arm/Group | Arm 1 Capecitabine and RT | Arm 2 Paclitaxel/Trastuzumab and RT | Arm 3: Paclitaxel and RT | Arm 4: Paclitaxel/Trastuzumab and RT
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm 1 Capecitabine and RT | Arm 2 Paclitaxel/Trastuzumab and RT | Arm 3: Paclitaxel and RT | Arm 4: Paclitaxel/Trastuzumab and RT
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No